CLINICAL TRIAL: NCT05743738
Title: Description of Septic Thrombophlebitis on Central Venous Catheter and Midline
Acronym: THROMBOSEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHM-2020/S10/14
Record Dates: First submitted 2023-02-10; First posted 2023-02-24 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-02

CONDITIONS: Septic Thrombophlebitis
Keywords: septic thrombophlebitis; Doppler ultrasound
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presence of thrombosis (Other): Doppler ultrasound D8, D15, D30, D45, D60 and D90
  Interventions: Diagnostic Test: Doppler ultrasound
- Absence of thrombosis (No Intervention)

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — Control venous Doppler ultrasound
  Arms: Presence of thrombosis

SUMMARY:
Central venous catheters improve the tolerability and feasibility of patient care in the hospital setting by allowing the administration of hyper-osmotic, vesicant and venotoxic fluids. Despite these advantages, the long-term presence of central venous catheters is associated with thrombotic and infectious risks , including catheter-related bacteremia, which can be complicated by septic thrombophlebitis and endocarditis that can lead to death.

Septic thrombophlebitis is a complication of venous catheter infections, which increases the morbidity. It is defined by the presence of a thrombosis in the vein where the venous catheter is located, associated with a bacteremia. A distinction is made between superficial and deep thrombophlebitis.

The frequency of septic thrombophlebitis of venous catheters is variable and poorly described in the literature.

When the diagnosis of septic thrombophlebitis is made, it is recommended to extend the duration of antibiotic therapy, to remove the infected catheter and to prescribe anticoagulant treatment. However, there is no recommendation on the duration of anticoagulation for septic thrombophlebitis, whether it is deep or superficial.

Investigator proposes a prospective and descriptive interventional study to describe the ultrasound evolution of thrombus in patients with septic thrombophlebitis on central venous catheter and midline.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalised at the CHM or CHUA, with a central venous device (Implantable chamber, central venous jugular, femoral, subclavian, PICCline, dialysis catheter) or a Midline and having catheter-related bacteremia
* Catheter-related bacteremia according to the following definition (ePOPI): Positive blood cultures within 48 hours of a suspected catheter infection (or its removal) With one of the following criteria: - Before catheter removal: differential time of positivity of central/peripheral blood cultures ≥ 2 hours
* After catheter removal: positive catheter culture ≥ 103 CFU/ml, with the same organism.
* Patient transportable for ultrasound or ultrasound can be performed in the patient's bed
* Patient capable of giving consent, or consent of the trusted person for patients not capable of giving consent at the time of inclusion
* Written consent signed by the participant and the investigator
* Person affiliated to social security

Exclusion Criteria:

* Patient with a life expectancy of less than one month
* Contraindication to anticoagulation
* Patient already on curative anticoagulant therapy for any indication
* Minor or adult patient under guardianship or protected or deprived of liberty
* Pregnant, nursing or parturient woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of duration of ultrasound signs of septic thrombophlebitis on central venous catheter and midline | Day 90
  the duration is measured by time from the day of diagnosis of septic thrombophlebitis to the day of disappearance of signs of thrombophlebitis on Doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Angers, Angers
  - Centre Hospitalier Le Mans, Le Mans

IPD SHARING:
Plan to Share IPD: No